CLINICAL TRIAL: NCT02892656
Title: Reliability and Responsiveness of the Danish Version of the Pain Self-Efficacy Questionnaire in Patients With Chronic Low Back Pain
Brief Title: Reliability and Responsiveness of One Questionnaire Used on a Low Back Pain Population
Status: Completed | Type: Observational
Sponsor: Sano (Other)
Responsible Party: Sponsor
Other Study IDs: Sano 2
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the reliability and responsiveness of the Pain Self-Efficacy Questionnaire (PSEQ) in a chronic low back pain (CLBP) population referred to The Danish Rheumatism Associations´ rehabilitation centre Sano Aarhus.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a highly prevalent health condition, and the leading cause of years lived with disability both globally and in Denmark. In the majority of patients with CLBP, no underlying pathology or cause can be identified and CLBP is acknowledged to be multifactorial. CLBP is defined by symptoms lasting for a period longer than three months. The high prevalence of CLBP causes a substantial impact on patients and their families, communities and health-care systems, as well as a financial burden. Besides pain and disability people with CLBP often experience psychosocial consequences with signs of anxiety and depression and effects on social, leisure, and work life.

An important component in rehabilitation is documentation of treatment outcomes. This demands that a change over time can be measured. To determine effect, the measurement tool must detect real or important change over time. This requires the measurement tool is reliable, and therefore will show no real or important change in periods where the patient is stable. If the measurement tool shows real or important change, in periods where there is no change in the patient state, the results can not be predicted as an effect from an intervention, but due to uncertainty of measurement tool.

The measurement tool is selected by the recommendation of literature and involvement of clinicians and patients at sano, and examines patient with CLBP.

It is found necessary to determine the reliability and responsiveness of the PSEQ on the CLBP population referred to Sano Aarhus. Data will be electronically entered in, stored in and collected from Sanos internal database (SanoBasen).

ELIGIBILITY:
Inclusion Criteria:

• referred to The Danish Rheumatism Associations' rehabilitation centre Sano

Exclusion criteria:

* a rated physical status of > 3 according to the American Society of Anesthesiologists Physical Status Classification System
* axial spondyloarthritis
* spinal fracture within the last 3 months
* severe osteoporosis
* active cancer
* active psychiatric pathology assessed by general practitioner before referral
* pregnancy
* low Danish language skills
* no e-mail address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain (defined as pain lasting for more than 12 months) with or without sciatica and/or with or without generalized pain identified by ICD-10 codes.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Pain Self-efficacy questionnaire | 12 months
  The PSEQ consists of 10 items, each item is scored on a seven-point Likert scale with responses ranging from 0 (not at all confident) to 6 (completely confident). A total score is calculated by summing the scores of the 10 items yielding a total sum score ranging from 0-60. Higher scores indicate a stronger self-efficacy belief

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mette Schmidt, Msc. H.S., Principal Investigator — Sano
Locations (2):
- Denmark (2):
  - Sano, Middelfart
  - Sano, Skælskør

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vejlgaard C, Maribo T, Riisgaard Laursen J, Schmidt AM. Reliability and smallest detectable change of the Danish version of the Pain Self-Efficacy Questionnaire in patients with chronic low back pain. Scand J Pain. 2021 Jun 2;21(4):809-813. doi: 10.1515/sjpain-2021-0014. Print 2021 Oct 26. PMID 34062626